CLINICAL TRIAL: NCT01090778
Title: Pharmacokinetic Profiles of GH Using Two Different Administration Regimes; a Bolus and an Infusion Both With and Without Exercise, in Adults With Growth Hormone Deficiency
Brief Title: Diurnal Variation of Exogenous Peptides (GH Puls/Jurgita I)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Jurgita Janukonyte, Medical doctor, Aarhus University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2010/0121
Record Dates: First submitted 2010-03-22; First posted 2010-03-23 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Growth Hormone Deficiency
Keywords: growth hormone deficiency; circadian variation
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Human Growth Hormone; Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Norditropin SimpleXx sc bolus injection (Other): Single sc bolus injection of 3 mg growth hormone without interval exercise
  Interventions: Drug: Norditropin SimpleXx (growth hormone)
- Norditropin SimpleXx single sc injection (Other): Single sc bolus injection of 3 mg growth hormone with interval exercise
  Interventions: Drug: Norditropin SimpleXx (growth hormone)
- Norditropin SimpleXx contin. sc infusion (Other): Continuous sc infusion of 3 mg growth hormone without interval exercise
  Interventions: Drug: Norditropin SimpleXx (growth hormone)
- Norditropin SimpleXx cont. sc infusion (Other): Continuous sc infusion of 3 mg growth hormone with interval exercise
  Interventions: Drug: Norditropin SimpleXx (growth hormone)

INTERVENTIONS:
Drug: Norditropin SimpleXx (growth hormone) — 3mg/subject/day over two consecutive days
  Other Names: Norditropin® SimpleXx®

SUMMARY:
This is an exploratory trial with four cross-over arms measuring the pharmacokinetic and pharmacodynamic profiles of growth hormone using two different modes of growth hormone administration (subcutaneous infusion into the abdomen or subcutaneous bolus injection in the thigh) in 8 adult male or female patients with growth hormone deficiency during interval exercise or in supine rest. The order of dosing regimen within the groups and between the groups will be randomised. All patients will go through four different treatment sessions:A/B Single subcutaneous bolus injection, supine rest without/with interval exercise, sessions C/D: Continuous subcutaneous infusion, supine rest without/with interval exercise. Hypotheses: 1) There is day-to-day variation of exogenous growth hormone, 2)Concentration of growth hormone decreases due to exercise compared to supine rest, 3)There is a circadian variation in pharmacokinetics of exogenous growth hormone infused subcutaneously

DETAILED DESCRIPTION:
The subjects will attend a screening visit and four treatment sessions. The dosing visits will comprise either 2-day hospital stay for the bolus injection group or 3 day hospital stay for the infusion group.

ELIGIBILITY:
Inclusion Criteria:

* AGHD male or female subjects
* Stable GH replacement therapy for at least 3 months
* Body Mass Index 18,5 to 35.0 kg/m2
* Achieved final height
* Age ≥ 18 years

Exclusion Criteria:

* Known or suspected allergy to trial product or components of the trial product
* Subjects with active malignancy
* Severe cardiac insufficiency classified according to NYHA III-IV
* Unstable angina pectoris, acute myocardial infarction within the last 12 months
* Severe, uncontrolled hypertension: sitting blood pressure > 180/110 mmHg
* HbA1C > 7,5 %
* Impaired kidney function: plasma creatinine ≥ 150 umol/l according to the hospital lab.
* Impaired liver function: liver parameters exceed 2 times or more the upper normal limit, according to the hospital lab.
* Patients on insulin treatment
* Stable pituitary replacement therapy for less than 3 months
* Participation in any other clinical trial involving any investigational products within the last three months prior to this trial
* Any diseases judged by the investigator that could affect the trial
* Women of fertile age, who are pregnant, planning to become pregnant or breast-feeding. Women of fertile age, who are not currently using adequate contraception methods such as: contraceptive pills, IUD or who had not undergone hysterectomy or sterilization

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic profiles of growth hormone | 48 hours
  Pharmacokinetic profiles of growth hormone administrated subcutaneously (3 mg/day) as a bolus in the adult patients with growth hormone deficiency during interval exercise or in supine rest.

SECONDARY OUTCOMES:
Pharmacokinetic profiles of growth hormone | 60 hours
  To compare pharmacokinetic profiles of growth hormone administrated subcutaneously (3 mg/day) as an infusion in the adult patients with growth hormone deficiency during interval exercise or in supine rest.

CONTACTS AND LOCATIONS:
Overall Officials: Torben Laursen, professor, Principal Investigator — Institute of Pharmacology, Aarhus University
Locations (2):
- Denmark (2):
  - Medical Department M, Aarhus University Hospital, Aarhus C, Central Jutland
  - Aarhus University Hospital, Aarhus C